CLINICAL TRIAL: NCT06033222
Title: Developing an Approach to Perturbation of Human Small Intestinal and Colonic Permeability in Healthy Participants
Brief Title: A Study of Perturbation of Human Small Intestinal Colonic Permeability
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 23-003520
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — ricinoleic acid

STUDY DESIGN:
Intervention Model Description: Prospective randomized, placebo-control study of effect of castor oil on intestinal and colonic permeability
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- 750 mg castor oil treatment group (Experimental): Subjects will take ricinoleic acid daily on an empty stomach in the morning 30 minutes before breakfast for a total of 4 days
  Interventions: Dietary Supplement: Ricinoleic Acid 750 mg
- 1500 mg castor oil treatment group (Experimental): Subjects will take ricinoleic acid daily on an empty stomach in the morning 30 minutes before breakfast for a total of 4 days
  Interventions: Dietary Supplement: Ricinoleic Acid 1500 mg
- 3000 mg castor oil treatment group (Experimental): Subjects will take ricinoleic acid daily on an empty stomach in the morning 30 minutes before breakfast for a total of 4 days
  Interventions: Dietary Supplement: Ricinoleic Acid 3000 mg
- Placebo group (Placebo Comparator): Subjects will take placebo daily on an empty stomach in the morning 30 minutes before breakfast for a total of 4 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Ricinoleic Acid 750 mg — 750 mg administered orally
  Arms: 750 mg castor oil treatment group
Dietary Supplement: Ricinoleic Acid 1500 mg — 1500 mg administered orally
  Arms: 1500 mg castor oil treatment group
Dietary Supplement: Ricinoleic Acid 3000 mg — 3000 mg administered orally
  Arms: 3000 mg castor oil treatment group
Drug: Placebo — Contains no active ingredient.
  Arms: Placebo group

SUMMARY:
The purpose of this study is to evaluate the effect of castor oil versus placebo on intestinal permeability in healthy individuals.

DETAILED DESCRIPTION:
Randomized, parallel-group, placebo-controlled, blinded, dose-response study using Castor oil and see the effects it has on small bowel and colonic permeability measured in healthy female and male adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-obese, non-pregnant volunteers.
* 1:1 Male/Female Ratio.
* BMI < 30 kg/m^2.

Exclusion Criteria:

* Diabetes.
* Uncontrolled hypertension (with BP measured > 140/90mmHg in the CRTU)
* BMI ≥ 30 kg/m^2.
* Chronic NSAID use (> 1 day/week).
* Use of oral antibiotics for 2 weeks prior to and during the entire 5 day study period.
* Known intolerance of castor oil.
* Diagnosis of gastrointestinal diseases that are associated with abnormal intestinal or colonic permeability such as inflammatory bowel diseases, irritable bowel syndrome and celiac disease.
* Prior intestinal or colonic resection.
* Participation in highly vigorous exercise such as running > 5 miles per day in week prior to the permeability test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in urinary excretion of 13^C-mannitol | 0-2 hours, 2-8 hours and 8-24 hours
  Percent urinary excretion of 13^C-mannitol

SECONDARY OUTCOMES:
Change in urinary excretion of lactulose | 0-2 hours, 2-8 hours and 8-24 hours
  Percent urinary excretion of lactulose

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No